CLINICAL TRIAL: NCT02901041
Title: Interdisciplinary Study of Two Novel Anticonvulsants in Alcoholism
Brief Title: Interdisciplinary Study of A Novel Anticonvulsant in Alcoholism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: Mclean Hospital (Other); University of Houston (Other)
Responsible Party: Principal Investigator, Todd Farchione, Research Associate Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2R01AA015923-06 (NIH)
Record Dates: First submitted 2016-08-29; First posted 2016-09-15 (Estimated); Results first posted 2023-05-06 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-05

CONDITIONS: Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — Zonisamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Zonisamide & Computerized Psychotherapy (Experimental): Zonisamide capsules (with a target maintenance dose of 400 mg daily) and a seven module computerized psychotherapy for alcohol use disorders called Take Control (9 sessions) will be administered over the course of 12 weeks, followed by a two week medication taper.
  Interventions: Drug: Zonisamide; Behavioral: Take Control
- Placebo & Computerized Psychotherapy (Active Comparator): Placebo capsules (for zonisamide) and a seven module computerized psychotherapy for alcohol use disorders called Take Control will be administered over the course of 14 weeks.
  Interventions: Behavioral: Take Control; Drug: Placebo (for Zonisamide)

INTERVENTIONS:
Drug: Zonisamide — ZONEGRAN® (zonisamide) is an antiseizure drug chemically classified as a sulfonamide and unrelated to other antiseizure agents. A dose of 400 mg daily will be used as the target maintenance dose in this study but dosing will be modified if needed to adjust for subject tolerance of drug dosing.
  Other Names: Zonegran
  Arms: Zonisamide & Computerized Psychotherapy
Behavioral: Take Control — Take Control is a seven module computer-based intervention which presents evidence-based alcohol education that includes motivational interviewing and cognitive-behavioral skills building. This program is derived from the National Institute on Alcohol Abuse and Alcoholism's (NIAAA's) self-help approach, Rethinking Drinking.
  Starting on March 23, 2020, participants will participate in a simplified Take Control treatment at home due to the COVID-19 pandemic
Drug: Placebo (for Zonisamide) — Sugar pills manufactured to mimic Zonisamide capsules.
  Arms: Placebo & Computerized Psychotherapy

SUMMARY:
Alcoholism is the third leading cause of preventable death in the US, accounting for 80,000 deaths annually. Almost 18 million US adults have alcohol use disorder (AUD); however, approved medications for the treatment of AUD has shown limited effectiveness.

Zonisamide (ZON), a broad spectrum anticonvulsant, has proven to be more effective than a placebo in reducing alcohol intake in individuals with alcohol dependence. ZON's mechanism of action seems to be quite distinct from currently approved anti-alcoholism medications, which holds promise for treatment of individuals who are not responsive to conventional medications. However, much remains unknown about ZON's therapeutic mechanisms and ZON's efficacy in treating patients with a diagnosis of AUD.

To fill in these gaps, the investigators will conduct a double-blind randomized controlled study that assesses ZON's treatment mechanisms and effectiveness in reducing alcohol consumption in patients with AUD. Participants will be randomized to one of two conditions: 1) treatment with ZON and a computerized psychotherapy platform called Take Control (TC); 2) treatment with a placebo (PLC) and TC. To understand the neurobiology behind ZON's potential therapeutic effects on AUD, fMRI will be used to compare the brain activity of the ZON+TC versus PLC+TC group while participants perform an alcohol and emotional-word Stroop task, as well as an alcohol related cues task.

DETAILED DESCRIPTION:
Potential participants will complete a telephone and an in-clinic screening to determine eligibility for this study. Eligible participants will be randomized to receive one of two treatment conditions: 1) Zonisamide plus Take Control (a computerized alcohol reduction and medication compliance program developed by the National Institute on Alcohol Abuse and Alcoholism (NIAAA)); 2) a placebo plus Take Control. For both conditions, participants will receive 12 treatment sessions. Participants will receive medication at each session, and they should have two weeks worth of medication on hand at any given time. Participants will take the medication as prescribed at home. The first 11 treatment sessions will include Take Control. The 12 treatment sessions will be followed by two drug dose taper sessions, and a follow up phone interview immediately following the final session.

Participants will also undergo two scans of less than 2 hours duration, one before they begin study sessions and the second near the end of the study (12th study week and before the medication taper). At the in-clinic screening session, participants will receive a "MRI Information for Research Participants" handout that answers some commonly asked questions about MRI and tells participants what they can expect while undergoing an MRI scan. Both scans will be conducted at BU CILSE. Participants will be screened before each scan session for pregnancy (urine sample, women of childbearing potential only), recent smoking or alcohol use (breathalyzers), and illicit substance use (urine sample). Participants will be asked to complete the Alcohol Urge Questionnaire (AUQ) before and after the scan. Eligible participants will complete a 1-hour 3 Tesla MRI scan involving structural imaging (MRI) and functional imaging (fMRI). The fMRI scans include a resting-state scan (no task involved) a cognitive (Stroop) task, and an alcohol cue reactivity task. The latter two scans involve presentation of visual images to participants while they are in the scanner. No contrast agent or invasive procedures are used. Only personnel trained in working in high magnetic field environments will work on this project. Imaging data will be analyzed on secure networks using only encrypted files. All data obtained will be coded to protect participant privacy and confidentiality.

Starting on March 23, 2020, all study procedures have been moved to HIPAA compliant, remote platforms and can be performed from home due to the COVID-19 pandemic. Screenings will take place over the phone or Zoom, neurocognitive assessments will take place on Inquisit 5 at sessions 1 and 12, female participants of child-bearing potential will be directed to take a pregnancy test at all sessions, and patients will use a breathalyzer provided by Boston University at the start of each session to show they are within study-specified limits of blood alcohol content.

One month following completion of study treatment (study week 16), participants will be asked to complete a follow-up telephone assessment.

The entire study is estimated to be completed in five years. The first six months to nine months of the project will be dedicated to hiring, training and certifying staff. Recruitment will begin within three months of obtaining IRB approval, during Year 1 of the study. Approximately 3-4 new participants will be recruited per month. We anticipate recruiting a total of 5 participants in Year 1, 25 participants in Years 2 and 3, 30 participants in year 4, and 15 participants in Year 5. The last third of Year 5 will be devoted to completion of data entry and data management procedures, preliminary analyses, and the preparation of manuscripts

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis of an Alcohol Use Disorder (AUD)
* Adults ages 21 to 65 years old
* Expressed desire to stop drinking alcohol completely or to reduce alcohol consumption
* Reported drinking an average of at least 14 standard drinks per week for males, or 7 for females occurring over a 28-consecutive day period during the 90 day-long time window that preceded the screening session
* Must be willing to discontinue psychotherapy for substance use disorder (except A.A.)

Exclusion Criteria:

* Bipolar disorder, schizophrenia, current bulimia/anorexia, dementia, or other substance use disorder, with the exception of nicotine, marijuana, and caffeine
* Clear and current suicidal risk
* Significant medical problem (e.g. uncontrolled diabetes)
* Medical contraindication to the use of ZON (e.g. history of significant renal disease, kidney stones, liver problems, metabolic acidosis, etc), as indicated by the FDA Zonisamide medication guide
* History of anticonvulsant-induced rash
* Currently taking:

  1. acamprosate, naltrexone, topiramate, disulfiram, or benzodiazepines
  2. a medication that is a moderate or major inhibitor or inducer of cytochrome P450 3A4 enzymes
  3. an amphetamine or other psychomotor stimulant
  4. opioids or have been treated chronically with opioids
  5. antipsychotic agents, anticonvulsants, or sedative hypnotics
  6. drugs with "sulfa" moiety (e.g. sulfonamides, sulfonylureas, carbonic anhydrase inhibitors, thiazides, and loop diuretics), except ethacrynic acid
  7. anxiolytics or antidepressants
* Previously received ZON for the treatment of an AUD
* Known allergy to sulfonamides
* Implantation of anything containing magnetically sensitive material including metal plates, aneurysm clips, and cardiac pacemakers, stents
* Non-English speakers
* Pregnant women or women who are lactating (breastfeeding)

Exclusion from Screening:

* Reduction in the mean number of drinks consumed per week for the pre-screening period by 50% or more during the screening period or report of average drinks per day fall within safe levels of alcohol consumption (i.e. 2 drinks/day for males and 1 drink/day for females by the HHS standard) two weeks prior to screening
* Women of child bearing potential (not postmenopausal for at least one year) will not be admitted into this study unless they are found to have a negative HCG test during screening. If they pass the HCG screening, they will be asked to maintain the use of an effective means of contraception during the course of the study
* Blood test shows lower than average red or white blood cell count or higher than average level of acid in blood

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H Barlow, PhD, Principal Investigator — Boston University
Locations (1):
- Center for Anxiety and Related Disorders - Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Zonisamide & Computerized Psychotherapy: Zonisamide capsules (with a target maintenance dose of 400 mg daily) and a seven module computerized psychotherapy for alcohol use disorders called Take Control (9 sessions) will be administered over the course of 12 weeks, followed by a two week medication taper.
  Zonisamide: ZONEGRAN® (zonisamide) is an antiseizure drug chemically classified as a sulfonamide and unrelated to other antiseizure agents. A dose of 400 mg daily will be used as the target maintenance dose in this study but dosing will be modified if needed to adjust for subject tolerance of drug dosing.
  Take Control: Take Control is a seven module computer-based intervention which presents evidence-based alcohol education that includes motivational interviewing and cognitive-behavioral skills building. This program is derived from the National Institute on Alcohol Abuse and Alcoholism's (NIAAA's) self-help approach, Rethinking Drinking.
  Starting on March 23, 2020, participants will participate in a simplified Take Control treatment at home due to the COVID-19 pandemic
- Placebo & Computerized Psychotherapy: Placebo capsules (for zonisamide) and a seven module computerized psychotherapy for alcohol use disorders called Take Control will be administered over the course of 14 weeks.
  Take Control: Take Control is a seven module computer-based intervention which presents evidence-based alcohol education that includes motivational interviewing and cognitive-behavioral skills building. This program is derived from the National Institute on Alcohol Abuse and Alcoholism's (NIAAA's) self-help approach, Rethinking Drinking.
  Starting on March 23, 2020, participants will participate in a simplified Take Control treatment at home due to the COVID-19 pandemic
  Placebo (for Zonisamide): Sugar pills manufactured to mimic Zonisamide capsules.
Period: Overall Study
Arm/Group | Zonisamide & Computerized Psychotherapy | Placebo & Computerized Psychotherapy
Started | 40 | 41
Completed | 29 | 30
Not Completed | 11 | 11
Not completed — Withdrawal by PI | 4 | 8
Not completed — Withdrawal by Subject | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zonisamide & Computerized Psychotherapy | Placebo & Computerized Psychotherapy | Total
Number analyzed (Participants) | 40 | 41 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 41 | 81
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.28 (12.61) | 40.39 (10.64) | 41.81 (11.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 9 | 26
  Male | 23 | 32 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 36 | 35 | 71
  Unknown or Not Reported | 3 | 6 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 35 | 37 | 72
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 40 | 41 | 81
Alcohol Use Disorder Clinical Severity Rating [Mean (Standard Deviation); unit: units on a scale] — Alcohol Use Disorder was assessed using the Anxiety and Related Disorders Interview Schedule for DSM-5 (ADIS-5). This semi-structured, diagnostic clinical interview focuses on a subset of DSM-5 diagnoses. Diagnoses are assigned a clinical severity rating (CSR) on a scale from 0 (no symptoms) to 8 (extremely severe symptoms), with a rating of 4 or above (definitely disturbing/disabling) passing the clinical threshold for DSM diagnostic criteria.
  units on a scale | 5.35 (0.92) | 5.02 (0.91) | 5.19 (0.92)

OUTCOME MEASURES:

1. Primary Outcome: Average Standard Drinking Units Per Day
Description: Timeline followback (TLFB) was used to collect information on participant's daily drinking. TLFB is a form of interview used to collect retroactive data related to participant's drinking. Participants are presented with a calendar are asked to report what they drank each day for a specified timeframe (e.g. in the past week). Participants were encouraged to give their best estimate in the absence of total certainty regarding their drinking on a given day. Study assessors then used these responses to identify how many standard drinking units participants drank each day. The National Institute of Alcohol Abuse and Alcoholism (NIAAA) defines "one standard drinking unit" as containing 14 grams of pure alcohol, and provide guidelines for calculating standard drinking units based on the alcohol content and size of a given drink. TLFB data from 28 days before BL were used to calculate pre-treatment outcomes. In instances where 28 days of data were not available, 21 days were used instead.
Time Frame: Pre-treatment
Population: All participants were assessed on this measure at baseline.
Measure: Mean (Standard Deviation); unit: standard drinking units per day
Arm/Group | Zonisamide & Computerized Psychotherapy | Placebo & Computerized Psychotherapy
Number analyzed (Participants) | 40 | 41
standard drinking units per day | 4.50 (3.89) | 4.48 (2.44)
Statistical Analysis 1: Comparison: Placebo & Computerized Psychotherapy; A t-test was used to compare means between conditions at baseline (pre-treatment). The null hypothesis was that the difference in group means is zero; Test type: Superiority; p = .98, t-test, 2 sided; t=0.03, df=79.00; Mean Difference (Net) = 0.02, 95% CI 2-sided [-1.41 to 1.45]

2. Primary Outcome: Average Standard Drinking Units Per Day
Description: as for outcome 1
Time Frame: Post-treatment (Week 12)
Population: Fewer participants were analyzed at post-treatment (compared to pre-treatment) due to participant drop-out.
Measure: Mean (Standard Deviation); unit: standard drinking units per day
Arm/Group | Zonisamide & Computerized Psychotherapy | Placebo & Computerized Psychotherapy
Number analyzed (Participants) | 29 | 29
standard drinking units per day | 2.23 (2.15) | 3.06 (1.99)
Statistical Analysis 1: Comparison: Placebo & Computerized Psychotherapy; A t-test was used to compare means between conditions at baseline post-treatment. The null hypothesis was that the difference in group means is zero; Test type: Superiority; p = .13, t-test, 2 sided; t=-1.52, df=56.00; Mean Difference (Net) = -0.83, 95% CI 2-sided [-1.92 to 0.26]

3. Primary Outcome: Percentage of Drinking Days
Description: as for outcome 1
Time Frame: Pre-treatment
Population: All participants were analyzed for this measure.
Measure: Mean (Standard Deviation); unit: Percentage of drinking days
Arm/Group | Zonisamide & Computerized Psychotherapy | Placebo & Computerized Psychotherapy
Number analyzed (Participants) | 40 | 41
Percentage of drinking days | 72.77 (26.13) | 79.62 (19.78)
Statistical Analysis 1: Comparison: Placebo & Computerized Psychotherapy; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .19, t-test, 2 sided — Equality of variance was not assumed; t=-1.33, df=72.65; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.17 to 0.03]

4. Primary Outcome: Percentage of Drinking Days
Description: as for outcome 1
Time Frame: Post-treatment (Week 12)
Population: Fewer participants were analyzed at post-treatment (compared to pre-treatment) due to participant drop-out.
Measure: Mean (Standard Deviation); unit: percentage of drinking days
Arm/Group | Zonisamide & Computerized Psychotherapy | Placebo & Computerized Psychotherapy
Number analyzed (Participants) | 29 | 29
percentage of drinking days | 51.27 (32.35) | 68.14 (32.24)
Statistical Analysis 1: Comparison: Placebo & Computerized Psychotherapy; Test type: Superiority; p = .05, t-test, 2 sided; t=-1.99, df=56.00; Mean Difference (Net) = -0.17, 95% CI 2-sided [-0.34 to 0.00]

5. Primary Outcome: Percent Heavy Drinking Days
Description: TLFB was be used to estimate participants' daily drinking. In this assessment, participants are presented with a calendar and asked to provide retrospective estimates of their daily alcohol consumption over a specified time period. TLFB was used to gather information on participants' daily drinking. In this assessment, participants are presented with a calendar and asked to provide retrospective estimates of their daily alcohol consumption over a specified time period. TLFB data from 28 days before BL were used to calculate pre-treatment outcomes. In instances where 28 days of data were not available, 21 days were used instead. Heavy drinking days refers to the percentage of heavy drinking days within that window (4 or more drinks for women, 5 or more for men).
Time Frame: Pre-treatment
Population: All participants were analyzed for this measure.
Measure: Mean (Standard Deviation); unit: percentage of heavy drinking days
Arm/Group | Zonisamide & Computerized Psychotherapy | Placebo & Computerized Psychotherapy
Number analyzed (Participants) | 40 | 41
percentage of heavy drinking days | 46.43 (30.86) | 43.82 (32.49)
Statistical Analysis 1: Comparison: Placebo & Computerized Psychotherapy; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .71, t-test, 2 sided; t=0.37,df=79.00; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.11 to 0.17]

6. Primary Outcome: Percent Heavy Drinking Days
Description: TLFB was be used to estimate participants' daily drinking. (See outcome measure 1 for more details description.) In this assessment, participants are presented with a calendar and asked to provide retrospective estimates of their daily alcohol consumption over a specified time period. TLFB data from 28 days before post-treatment were used to calculate post-treatment outcomes. In instances where 28 days of data were not available, 21 days were used instead. Heavy drinking days refers to the percentage of heavy drinking days within that window (4 or more drinks for women, 5 or more for men).
Time Frame: Post-treatment (Week 12)
Population: Fewer participants were analyzed at post-treatment (compared to pre-treatment) due to participant drop-out.
Measure: Mean (Standard Deviation); unit: Percent heavy drinking days
Arm/Group | Zonisamide & Computerized Psychotherapy | Placebo & Computerized Psychotherapy
Number analyzed (Participants) | 29 | 29
Percent heavy drinking days | 19.83 (23.22) | 31.12 (30.38)
Statistical Analysis 1: Comparison: Placebo & Computerized Psychotherapy; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .12, t-test, 2 sided; t=-1.59,df=56.00; Mean Difference (Net) = -0.11, 95% CI 2-sided [-0.26 to 0.03]

7. Primary Outcome: Average Weekly Standard Drinking Units (SDUs)
Description: Timeline follow back is a form of interview used to collect retroactive data related to participant's drinking. Participants are presented with a calendar are asked to report what they drank each day for a specified timeframe (e.g. in the past week). Participants were encouraged to give their best estimate in the absence of total certainty regarding their drinking on a given day. Study assessors then used these responses to identify how many standard drinking units participants drank each day. The National Institute of Alcohol Abuse and Alcoholism (NIAAA) defines "one standard drinking unit" as containing 14 grams of pure alcohol, and provide guidelines for calculating standard drinking units based on the alcohol content and size of a given drink. These standards, which can be found the NIAAA website, were used to calculate participant's average drinking units.
Time Frame: Pre-treatment
Population: All participants were analyzed for this measure.
Measure: Mean (Standard Deviation); unit: standard drinking units per week
Arm/Group | Zonisamide & Computerized Psychotherapy | Placebo & Computerized Psychotherapy
Number analyzed (Participants) | 40 | 41
standard drinking units per week | 31.51 (27.23) | 31.37 (17.11)
Statistical Analysis 1: Comparison: Placebo & Computerized Psychotherapy; Test type: Superiority; p = .98, t-test, 2 sided; t=0.03, df=79.00; Mean Difference (Net) = 0.14, 95% CI 2-sided [-9.89 to 10.18]

8. Primary Outcome: Average Weekly Standard Drinking Units (SDUs)
Description: as for outcome 1
Time Frame: Post-treatment (Week 12)
Population: Fewer participants were analyzed at post-treatment (compared to pre-treatment) due to participant drop-out.
Measure: Mean (Standard Deviation); unit: standard drinking units per week
Arm/Group | Zonisamide & Computerized Psychotherapy | Placebo & Computerized Psychotherapy
Number analyzed (Participants) | 29 | 29
standard drinking units per week | 15.64 (15.03) | 21.43 (13.96)
Statistical Analysis 1: Comparison: Placebo & Computerized Psychotherapy; Test type: Superiority; p = .13, t-test, 2 sided; t=-1.52, df=56.00; Mean Difference (Net) = -5.80, 95% CI 2-sided [-13.43 to 1.83]

9. Secondary Outcome: Balloon Analogue Risk Task: Total Pump Count
Description: In this online task, participants are presented with a balloon. Clicking a button will pump the balloon, causing it to inflate and the participant to be awarded a certain amount of money. This happens until a threshold when a pump will cause the balloon to explode and all money would be lost. At any point in time, participants can choose between pumping the balloon further and risking it exploding, or not pumping the balloon and collecting the money they have already earned. 90 trials are conducted and the average number of pumps delivered are used to measure levels of risk-taking. Higher numbers of balloon pumps are associated with greater risk-taking.
Time Frame: Pre-treatment
Population: Not all participants completed the neurocognitive tests associated with the study.
Measure: Mean (Standard Deviation); unit: pumps
Arm/Group | Zonisamide & Computerized Psychotherapy | Placebo & Computerized Psychotherapy
Number analyzed (Participants) | 31 | 32
pumps | 709.23 (370.01) | 682.16 (307.33)
Statistical Analysis 1: Comparison: Placebo & Computerized Psychotherapy; Test type: Superiority; p = .75, t-test, 2 sided; t=0.32,df=61.00; Mean Difference (Net) = 27.07, 95% CI 2-sided [-144.06 to 198.20]

10. Secondary Outcome: Balloon Analogue Risk Task: Total Pump Count
Description: as for outcome 9
Time Frame: Post-treatment (Week 12)
Population: Fewer participants were analyzed at post-treatment (compared to pre-treatment) due to participant drop-out.
Measure: Mean (Standard Deviation); unit: pumps
Arm/Group | Zonisamide & Computerized Psychotherapy | Placebo & Computerized Psychotherapy
Number analyzed (Participants) | 22 | 26
pumps | 829.09 (409.84) | 730.04 (312.94)
Statistical Analysis 1: Comparison: Placebo & Computerized Psychotherapy; Test type: Superiority; p = .35, t-test, 2 sided; t=0.95, df=46.00; Mean Difference (Net) = 99.05, 95% CI 2-sided [-111.11 to 309.21]

11. Secondary Outcome: Cued Go/No-go Task: Inhibition Error
Description: In this online task, participants are first presented with a go or a no-go cue, and are then presented with a go or no-go target. Participants are instructed to respond to a go target by clicking on a button, and not to respond to a no-go target. The cues have a high probability of signaling a correct target (valid cues), and a low probability of signaling an incorrect target (invalid cues). Incorrect responses to the no-go target are used to assess inhibitory control, which reflect impulse control. A test includes 250 trials and takes approximately 15 minutes to complete. Here, inhibition error is reported as the error rate (as a percentage) for trials where a go cue was followed by a no-go target. Larger error rates reflect less inhibitory control.
Time Frame: Pre-treatment
Population: Not all participants completed the neurocognitive tests associated with the study.
Measure: Mean (Standard Deviation); unit: percentage of incorrect responses
Arm/Group | Zonisamide & Computerized Psychotherapy | Placebo & Computerized Psychotherapy
Number analyzed (Participants) | 28 | 32
percentage of incorrect responses | 2.48 (6.43) | 1.63 (3.02)
Statistical Analysis 1: Comparison: Placebo & Computerized Psychotherapy; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .51, t-test, 2 sided; t=0.67, df=58.00; Mean Difference (Net) = 0.85, 95% CI 2-sided [-1.69 to 3.40]

12. Secondary Outcome: Cued Go No-Go: Inhibition Error
Description: as for outcome 11
Time Frame: Post-treatment (Week 12)
Population: Fewer participants were analyzed at post-treatment (compared to pre-treatment) due to participant drop-out. One participant was excluded from the analyses due to highly elevated error rates (>80%).
Measure: Mean (Standard Deviation); unit: percentage of incorrect responses
Arm/Group | Zonisamide & Computerized Psychotherapy | Placebo & Computerized Psychotherapy
Number analyzed (Participants) | 19 | 19
percentage of incorrect responses | 0.63 (1.50) | 1.05 (2.61)
Statistical Analysis 1: Comparison: Placebo & Computerized Psychotherapy; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .55, t-test, 2 sided; t=-0.61,df=36; Mean Difference (Net) = -0.42, 95% CI 2-sided [-1.82 to 0.98]

13. Secondary Outcome: Connor's Continuous Performance Task (CPT) - X Test Omission Rate
Description: The CPT includes two attention tasks, the second one being more difficult than the first. In the first task (reported on here), participants are presented a series of letters, one letter by one letter, and are asked to click on a button when the letter X appears. The letters appear at approximately 0.92s intervals, and responses are scored correctly if the button is clicked within 0.69s after the letter appears. An omission occurs when the X appears but the participant does not click the button within 0.69 seconds after it appears. The omission rate is calculated by dividing the number of omissions by the number of X presentations and converting that to a percentage. Higher omission rates indicate worse performance on this attentional task.
Time Frame: Pre-treatment
Population: Not all participants completed the neurocognitive tests associated with the study. Two participants were excluded from the analyses due to highly elevated error rates (>80%)
Measure: Mean (Standard Deviation); unit: percentage of omitted responses
Arm/Group | Zonisamide & Computerized Psychotherapy | Placebo & Computerized Psychotherapy
Number analyzed (Participants) | 28 | 32
percentage of omitted responses | 23.51 (8.42) | 23.37 (8.20)
Statistical Analysis 1: Comparison: Placebo & Computerized Psychotherapy; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .95, t-test, 2 sided; t=0.07,df=58.00; Mean Difference (Net) = 0.15, 95% CI 2-sided [-4.15 to 4.45]

14. Secondary Outcome: Connor's Continuous Performance Task (CPT): X Test Omission Rate
Description: as for outcome 13
Time Frame: Post-treatment (Week 12)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: percentage of omitted responses
Arm/Group | Zonisamide & Computerized Psychotherapy | Placebo & Computerized Psychotherapy
Number analyzed (Participants) | 18 | 22
percentage of omitted responses | 29.76 (16.58) | 26.42 (8.76)
Statistical Analysis 1: Comparison: Placebo & Computerized Psychotherapy; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .42, t-test, 2 sided; t=0.82, df=38.00; Mean Difference (Net) = 3.34, 95% CI 2-sided [-4.93 to 11.62]

15. Secondary Outcome: Connor's Continuous Performance Task (CPT): X Test Commission Rate
Description: The CPT includes two attention tasks, the second one being more difficult than the first. In the first task (reported on here), participants are presented a series of letters, one letter by one letter, and are asked to click on a button when the letter X appears. The letters appear at approximately 0.92s intervals, and responses are scored correctly if the button is clicked within 0.69s after the letter appears. A commission occurs when a participant clicks a button when something other than the letter X has been presented. The commission rate is calculated by dividing the number of commissions by the total number of non-X presentations and converting that to a percentage. Higher commission rates indicate worse performance on this attentional task.
Time Frame: Pre-treatment
Population: Not all participants completed the neurocognitive tests associated with the study.
Measure: Mean (Standard Deviation); unit: percentage of commission responses
Arm/Group | Zonisamide & Computerized Psychotherapy | Placebo & Computerized Psychotherapy
Number analyzed (Participants) | 30 | 32
percentage of commission responses | 0.74 (1.20) | 0.42 (0.45)
Statistical Analysis 1: Comparison: Placebo & Computerized Psychotherapy; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .17, t-test, 2 sided — Equal variance was not assumed; t=1.39, df=36.37; Mean Difference (Net) = 0.32, 95% CI 2-sided [-0.15 to 0.80]

16. Secondary Outcome: Connor's Continuous Performance Task (CPT): X Test Commission Rate
Description: The CPT includes two attention tasks, the second one being more difficult than the first. In the first task (reported on here), participants are presented a series of letters, one letter by one letter, and are asked to click on a button when the letter X appears.The letters appear at approximately 0.92s intervals, and responses are scored correctly if the button is clicked within 0.69s after the letter appears. A commission occurs when a participant clicks a button when something other than the letter X has been presented. The commission rate is calculated by dividing the number of commissions by the total number of non-X presentations and converting that to a percentage. Higher commission rates indicate worse performance on this attentional task.
Time Frame: Post-treatment (Week 12)
Population: Fewer participants were analyzed at post-treatment (compared to pre-treatment) due to participant drop-out.
Measure: Mean (Standard Deviation); unit: percentage of commission responses
Arm/Group | Zonisamide & Computerized Psychotherapy | Placebo & Computerized Psychotherapy
Number analyzed (Participants) | 19 | 22
percentage of commission responses | 0.84 (1.09) | 0.43 (0.48)
Statistical Analysis 1: Comparison: Placebo & Computerized Psychotherapy; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.14, t-test, 2 sided — Equal variances were not assumed when conducting the t-test; t=1.53, df=24.05; Mean Difference (Net) = 0.41, 95% CI 2-sided [-0.14 to 0.97]

17. Secondary Outcome: Connor's Continuous Performance Task (CPT): AX Test Omission Rate
Description: The CPT includes two attention tasks, the second one being more difficult than the first. In the second task (reported on here), participants are presented with a series of letters, and are instructed to click on the button only when the letter X appears directly after the letter A appears (an AX presentation). The letters appear at approximately 0.92s intervals, and responses are scored correctly if the button is clicked within 0.69s after the letter appears. An omission occurs when a participant does not click the button when the letter X appears directly after the letter A. The omission rate is calculated by dividing the number of omissions by the total number of AX presentations and converting that to a percentage. Higher omission rates indicate worse performance on this attentional task.
Time Frame: Pre-treatment
Population: Not all participants completed the neurocognitive tests associated with the study. One participant was excluded from the analyses due to highly elevated error rates (>80%).
Measure: Mean (Standard Deviation); unit: percentage of omission responses
Arm/Group | Zonisamide & Computerized Psychotherapy | Placebo & Computerized Psychotherapy
Number analyzed (Participants) | 29 | 32
percentage of omission responses | 6.40 (9.92) | 3.33 (4.76)
Statistical Analysis 1: Comparison: Placebo & Computerized Psychotherapy; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .14, t-test, 2 sided — Equal variances were not assumed when conducting the t-tests; t=1.51,df=39.34; Mean Difference (Net) = 3.07, 95% CI 2-sided [-1.03 to 7.16]

18. Secondary Outcome: Connor's Continuous Performance Task (CPT): AX Test Omission Rate
Description: The CPT includes two attention tasks, the second one being more difficult than the first. In the first task, participants are presented a series of 31 letters, one letter by one letter, and are asked to click on a button when the letter X appears. In the second task (reported on here), participants are presented with a series of 31 letters, and are instructed to click on the button only when the letter X appears directly after the letter A appears (an AX presentation). The letters appear at approximately 0.92s intervals, and responses are scored correctly if the button is clicked within 0.69s after the letter appears. An omission occurs when a participant does not click the button when the letter X appears directly after the letter A. The omission rate is calculated by dividing the number of omissions by the total number of AX presentations and converting that to a percentage. Higher omission rates indicate worse performance on this attentional task.
Time Frame: Post-treatment (Week 12)
Population: Fewer participants were analyzed at post-treatment (compared to pre-treatment) due to participant drop-out.
Measure: Mean (Standard Deviation); unit: percentage of omission responses
Arm/Group | Zonisamide & Computerized Psychotherapy | Placebo & Computerized Psychotherapy
Number analyzed (Participants) | 19 | 22
percentage of omission responses | 8.76 (13.99) | 5.58 (9.88)
Statistical Analysis 1: Comparison: Placebo & Computerized Psychotherapy; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .40, t-test, 2 sided — Equality of variance was not assumed; t=0.85, df=39.00; Mean Difference (Net) = 3.18, 95% CI 2-sided [-4.39 to 10.75]

19. Secondary Outcome: Connor's Continous Performance Task: AX Test Commission Rate
Description: The CPT includes two attention tasks, the second one being more difficult than the first. In the second task (reported on here), participants are presented with a series of letters, and are instructed to click on the button only when the letter X appears directly after the letter A appears (an AX presentation). The letters appear at approximately 0.92s intervals, and responses are scored correctly if the button is clicked within 0.69s after the letter appears. A commission occurs when a participant presses the button at any time other than following an AX presentation (i.e. during a non-AX presentation). The commission rate is calculated by dividing the number of commissions by the number of non-AX presentations and converting that to a percentage. Higher commission rates indicate worse performance on this attentional task.
Time Frame: Pre-treatment
Population: Not all participants completed the neurocognitive tests associated with the study.
Measure: Mean (Standard Deviation); unit: percentage of commission responses
Arm/Group | Zonisamide & Computerized Psychotherapy | Placebo & Computerized Psychotherapy
Number analyzed (Participants) | 30 | 32
percentage of commission responses | .80 (1.03) | 0.40 (0.43)
Statistical Analysis 1: Comparison: Placebo & Computerized Psychotherapy; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .06, t-test, 2 sided — Equal variances were not assumed when conducting the t-test; t=1.97, df=38.37; Mean Difference (Net) = .40, 95% CI 2-sided [-0.01 to 0.81]

20. Secondary Outcome: Connor's Continuous Performance Task: AX Test Commission Rate
Description: as for outcome 19
Time Frame: Post-treatment (Week 12)
Population: Fewer participants were analyzed at post-treatment (compared to pre-treatment) due to participant drop-out.
Measure: Mean (Standard Deviation); unit: percentage of commission responses
Arm/Group | Zonisamide & Computerized Psychotherapy | Placebo & Computerized Psychotherapy
Number analyzed (Participants) | 19 | 22
percentage of commission responses | 0.87 (1.65) | 0.84 (1.59)
Statistical Analysis 1: Comparison: Placebo & Computerized Psychotherapy; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .96, t-test, 2 sided; t=.06, df=39.00; Mean Difference (Net) = .03, 95% CI 2-sided [-1.00 to 1.05]

21. Secondary Outcome: Roger's Risk Task: Mean Percent Bet
Description: Participants are given 10 boxes. Some of these boxes are red, the others are blue. They are told that a yellow token is hidden under one of these boxes and they have to guess the color of the box under which the yellow token is hidden. Once they decide on the color, they are asked to bet points on this choice: the computer provides the bets in either ascending (bets get bigger) or descending order (bets get smaller) and participants are asked to click on a bet when they want to bet this number of points. If they win, the bet number is added to their total points. If they lose the bet number is taken away from their total points. "Mean percent bet" refers to the overall mean percentage of their points participants bet across trials.
Time Frame: Pre-treatment
Population: Not all participants completed the neurocognitive tests associated with the study.
Measure: Mean (Standard Deviation); unit: percentage of points bet
Arm/Group | Zonisamide & Computerized Psychotherapy | Placebo & Computerized Psychotherapy
Number analyzed (Participants) | 28 | 31
percentage of points bet | 61.51 (14.18) | 59.48 (14.93)
Statistical Analysis 1: Comparison: Placebo & Computerized Psychotherapy; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .60, t-test, 2 sided; t=0.53,df=57.00; Mean Difference (Net) = 2.03, 95% CI 2-sided [-5.58 to 9.64]

22. Secondary Outcome: Roger's Risk Task: Mean Percent Bet
Description: as for outcome 21
Time Frame: Post-treatment (Week 12)
Population: The number of participants analyzed at pre-treatment exceeds the number of participants analyzed at post-treatment due to participant dropout.
Measure: Mean (Standard Deviation); unit: percentage of points bet
Arm/Group | Zonisamide & Computerized Psychotherapy | Placebo & Computerized Psychotherapy
Number analyzed (Participants) | 19 | 22
percentage of points bet | 56.01 (15.28) | 61.62 (13.07)
Statistical Analysis 1: Comparison: Placebo & Computerized Psychotherapy; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .21, t-test, 2 sided; t=-1.27, df=39.00; Mean Difference (Net) = -0.06, 95% CI 2-sided [-0.15 to 0.03]

23. Secondary Outcome: Roger's Risk Task: Risk Adjustment
Description: Participants are given 10 boxes. Some of these boxes are red, the others are blue. They are told that a yellow token is hidden under one of these boxes and they have to guess the color of the box under which the yellow token is hidden. Once they decide on the color, they are asked to bet points on this choice: the computer provides the bets in either ascending (bets get bigger) or descending order (bets get smaller) and participants are asked to click on a bet when they want to bet this number of points. If they win, the bet number is added to their total points. If they lose the bet number is taken away from their total points. Risk adjustment is a measure of the difference between their risk taking behavior during ascending versus descending trials, and represents whether the participant changes their bet based on the odds of winning. There are no min or max scores, and a higher score indicates the subject is more likely to change the wager depending on the probability of winning.
Time Frame: Pre-treatment
Population: Not all participants completed the neurocognitive tests associated with the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Zonisamide & Computerized Psychotherapy | Placebo & Computerized Psychotherapy
Number analyzed (Participants) | 28 | 31
score on a scale | 0.67 (0.66) | 0.94 (0.57)
Statistical Analysis 1: Comparison: Placebo & Computerized Psychotherapy; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .09, t-test, 2 sided; t=-1.74,df=57.00; Mean Difference (Net) = -0.28, 95% CI 2-sided [-0.60 to 0.04]

24. Secondary Outcome: Roger's Risk Task: Risk Adjustment
Description: as for outcome 23
Time Frame: Post-treatment (Week 12)
Population: Fewer participants were analyzed at post-treatment (compared to pre-treatment) due to participant drop-out.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Zonisamide & Computerized Psychotherapy | Placebo & Computerized Psychotherapy
Number analyzed (Participants) | 19 | 22
score on a scale | 0.55 (0.74) | 0.91 (0.61)
Statistical Analysis 1: Comparison: Placebo & Computerized Psychotherapy; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .10, t-test, 2 sided; t=-1.69, df=39.00; Mean Difference (Net) = -0.35, 95% CI 2-sided [-0.78 to 0.07]

25. Secondary Outcome: Roger's Risk Task: Delay Aversion
Description: Participants are given 10 boxes. Some of these boxes are red, the others are blue. They are told that a yellow token is hidden under one of these boxes and they have to guess the color of the box under which the yellow token is hidden. Once they decide on the color, they are asked to bet points on this choice: the computer provides the bets in either ascending (bets get bigger) or descending order (bets get smaller) and participants are asked to click on a bet when they want to bet this number of points. If they win, the bet number is added to their total points. If they lose the bet number is taken away from their total points. Delay aversion is the difference between the risk-taking score in the descend and ascend conditions. There is no min or max score. Participants who find delays aversive tend to select an amount to bet early in the sequence; i.e., a large bet in the descend condition, and a small bet in the ascend condition. Thus, they will have a higher risk aversion score.
Time Frame: Pre-treatment
Population: Not all participants completed the neurocognitive tests associated with the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Zonisamide & Computerized Psychotherapy | Placebo & Computerized Psychotherapy
Number analyzed (Participants) | 28 | 31
score on a scale | 0.32 (0.34) | 0.30 (0.29)
Statistical Analysis 1: Comparison: Placebo & Computerized Psychotherapy; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.80, t-test, 2 sided; t=0.25,df=57.00; Mean Difference (Net) = 0.02, 95% CI 2-sided [-0.15 to 0.19]

26. Secondary Outcome: Roger's Risk Task: Delay Aversion
Description: as for outcome 25
Time Frame: Post-treatment (Week 12)
Population: Fewer participants were analyzed at post-treatment (compared to pre-treatment) due to participant drop-out.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Zonisamide & Computerized Psychotherapy | Placebo & Computerized Psychotherapy
Number analyzed (Participants) | 19 | 22
score on a scale | 0.16 (0.60) | 0.30 (0.42)
Statistical Analysis 1: Comparison: Placebo & Computerized Psychotherapy; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .41, t-test, 2 sided; t=-0.84,df=39.00; Mean Difference (Net) = -5.61, 95% CI 2-sided [-14.56 to 3.34]

ADVERSE EVENTS:
Time Frame: 14 weeks
Description: Serious adverse events were those that required immediate reporting to Boston University's Institutional Review Board according to their definitions of SAEs. All other adverse events were collected using the Modified SAFTEE form, administered by study physicians on a weekly basis. Percentages reflect the percent of participants who endorsed a given adverse event at any time during the trial.
Arm/Group | Zonisamide & Computerized Psychotherapy | Placebo & Computerized Psychotherapy
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/41
Serious Adverse Events (participants affected / at risk) | 2/40 | 1/41
Other Adverse Events (participants affected / at risk) | 20/40 | 20/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zonisamide & Computerized Psychotherapy (N=40) | Placebo & Computerized Psychotherapy (N=41)
Metabolic acidosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Episodic heart fluttering (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zonisamide & Computerized Psychotherapy (N=40) | Placebo & Computerized Psychotherapy (N=41)
Nausea (General disorders) | 3 (5) | 0 (0)
Decreased appetite (Gastrointestinal disorders) | 3 (6) | 1 (1)
Weight loss (General disorders) | 4 (9) | 3 (4)
Headache (General disorders) | 11 (22) | 5 (5)
Dizziness/Fainting (General disorders) | 3 (3) | 6 (7)
Nervousness/anxiety (Psychiatric disorders) | 2 (21) | 4 (10)
Memory problems (Psychiatric disorders) | 2 (2) | 1 (2)
Insomnia (Psychiatric disorders) | 5 (13) | 6 (11)
Drowsiness (General disorders) | 0 (0) | 4 (4)
Tiredness/Fatigue (General disorders) | 3 (11) | 5 (17)
Cough (General disorders) | 1 (1) | 3 (3)
Diarrhea (General disorders) | 3 (3) | 1 (2)
Dry mouth (General disorders) | 2 (2) | 0 (0)
Taste change (General disorders) | 5 (6) | 0 (0)
Fever (General disorders) | 2 (2) | 0 (0)
Congestion (General disorders) | 3 (5) | 4 (5)
Depression (Psychiatric disorders) | 2 (20) | 1 (12)
Concentration difficulties (Psychiatric disorders) | 2 (6) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-14): https://cdn.clinicaltrials.gov/large-docs/41/NCT02901041/Prot_SAP_001.pdf